CLINICAL TRIAL: NCT02534051
Title: A Clinical Care Pathway for Obese Pregnant Women: A Pilot Cluster Randomized Controlled Trial
Brief Title: A Clinical Care Pathway for Obese Pregnant Women: A Pilot Cluster RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Sarah McDonald, Principal Investigator, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Carepath
Record Dates: First submitted 2015-08-21; First posted 2015-08-27 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Obesity; Pregnancy
Keywords: clinical care path; care pathway; obesity; pregnancy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical care pathway (Active Comparator): The intervention is the clinical care pathway designed by investigators, informed by the national guideline co-authored by one of the team, and supplemented by the review of the literature
  Interventions: Other: Clinical Care Pathway
- Usual Care (No Intervention): The control group will receive the usual prenatal care.

INTERVENTIONS:
Other: Clinical Care Pathway — The clinical care pathway guides aspects of care specific to obese pregnant women:1st trimester: offer of testing for pre-existing diabetes with either 75g OGTT or 50g GCT, nuchal translucency ultrasound (u/s), calculation of body mass index, counselling about weight gain, advising about medical complications, screening for obstructive sleep apnea, and referral to Maternal-Fetal Medicine if history of bariatric surgery, 2nd trimester: offer of maternal-serum alpha fetal protein (spina bifida), anatomy u/s, and 50g GCT and 75g OGTT, 3rd trimester: offer of consultation with anesthesiology, u/s for growth & well-being, counselling about birth risks, and discussion of breastfeeding.
  Arms: Clinical care pathway

SUMMARY:
Clinics will be randomized to the use of the care pathway for obese pregnant women or standard care. Women who are (1) up to 20 weeks + 6 days gestation into their pregnancy, (2) are carrying one baby (not twins) that is healthy (no life threatening anomalies) and (3) have a Body Mass Index ≥ 30 kg/m², will be included. Data will be obtained from the Ministry of Health's Antenatal Records, charts, and for those in the intervention group, the care path (filled out by the practitioners - the participants' obstetrician, midwife, or family doctor). At the end of the study, practitioners will complete a survey, participate in structured interviews to understand barriers, facilitators, and motivators of using the care path.

Primary Objective:

To evaluate the feasibility of implementing and testing a clinical care pathway for obese pregnant women in a pilot cluster randomized controlled trial (RCT)

Secondary Objectives:

To obtain pilot data on A) process outcomes (steps of the pathway, e.g. what % of obese women receive a screen for diabetes) B) clinical outcomes (e.g. what % of obese women receive a diagnosis of diabetes), C) provider outcomes (e.g. Is the intervention acceptable, feasible & efficient? Barriers & facilitators to use, effectiveness? [Structured interviews])

DETAILED DESCRIPTION:
STUDY DESIGN:

Investigators propose a pilot cluster RCT with a 1:1 allocation ratio of clinics randomized to the clinical care pathway for obese pregnant women (intervention group) versus standard care (control group).

Investigators have followed the SPIRIT statement (Standard Protocol Items: Recommendations for Interventional Trials)

RANDOMIZATION:

The unit of randomization will be the clinic providing pregnancy care. All pregnant women who meet inclusion criteria at a clinic randomized to the intervention will receive the intervention, while all pregnant women who meet the inclusion criteria at a clinic randomized to usual care will receive usual care. Investigators used a 1:1 allocation between the intervention and the control groups, with paired randomization by type of clinic (obstetrician-lead versus midwife-lead, since they likely differ regarding patient characteristics and health care, and pairing will aid in providing a reasonable balance of characteristics with a small sample size.) Investigators generated the randomization sequence using www.randomization.com. The randomization seed for obstetrical clinics was "21262" and the randomization seed for midwifery clinics was "23340".

STUDY PROCESS:

Clinics will be randomly allocated to the intervention or control group, in a paired fashion (so that one of the two midwifery clinics is randomized to the intervention group and the other to the control, given that both the clinical care and the women in the clinics are more likely to be similar between these two clinics).

As the study involves a minimal/no-risk intervention, the Hamilton Integrated Research Ethics Board (HiREB) has approved clinics to be randomized and all eligible women at intervention clinics to receive the intervention (and all eligible women at control clinics to receive routine care); given that the intervention is standard of care, individual participant consent is not required. Informed, written consent of staff at the clinics which will be randomized to the intervention will be obtained prior to semi-structured interviews at the end of the study. Investigators do not plan an interim analysis given the minimal/no-risk nature of the intervention, and the pilot nature of the study, and hence investigators will not have a Data Safety Monitoring Board (DSMB), but will have a Steering Commitee.

DATA COLLECTION:

Data will be collected at the end of pregnancy from the:

1. 2-page Antenatal Records mandated by the Ministry of Health: baseline characteristics*, clinical and process outcomes
2. clinical care path (in intervention group): feasibility
3. clinic and hospital charts: process and clinical outcomes
4. care provider survey and structured interviews (in intervention group): provider outcomes.

   * Baseline characteristics will include: maternal age, education level, pre-existing diabetes or hypertension or other co-morbidities, gestational age upon first visit to randomized clinic, pre-pregnancy body mass index, gravidity, and parity.

SAMPLE SIZE:

Investigators have provided a sample size justification, rather than a calculation for the following reasons:

1. 'In general, sample size calculations may not be required for some pilot studies'
2. Given that this is a feasibility study, it was not designed to have statistical power to detect a difference between the 2 treatment groups.
3. The size of the intraclass correlation coefficient (ICC) required for a sample size calculation is currently unknown.

The sample size was based on feasibility considerations as follows: Investigators conservatively estimate there would be a total of 142 participants available (71 per group) over 10 months of recruitment, at 8 clinics, with 80% of women in the intervention clinics receiving the intervention, (and 100% of women in the control group receiving usual care), a variable rate of obesity from 20-30% depending on the clinic, and a variable proportion of women presenting to the clinic for prenatal care at <20 weeks+6 days gestation ranging from 15% in obstetrician-lead clinics to 85% in midwifery-lead clinics).

This number of patients, 71 per group, exceeds one common number for a sample size for a pilot study, the "of at least 50 per group", since additional power is required for cluster designs.

STATISTICAL ANALYSES:

Baseline characteristics and co-morbid conditions will be compared between women receiving the intervention versus those in the control group. Since the design of the study involves paired randomization, hence paired analysis will be performed. Continuous data will be compared using a paired t test for means (standard deviations) or Wilcoxon test for paired medians (interquartile range), as appropriate. Paired proportions for categorical variables will be compared using a McNemar's test.

The analysis of the primary outcome, feasibility, will be based on descriptive statistics of the proportions (%) of women in the intervention group who have the care path completed, and for whom care providers would recommend it. Analysis will be done at the patient level with the exception of care provider outcomes. Investigators will use intention to treat analysis, i.e. outcomes of all eligible women at the intervention clinic will be evaluated within the intervention group whether she received the intervention or not.

The analysis of the secondary outcomes (process outcomes and clinical outcomes) will be done using McNemar's test to compare paired proportions of women in the intervention group who receive the recommended care to the proportion of women in the control group who do.

Investigators will perform sensitivity analyses: 1) "per-protocol analysis", i.e. per-clinical care path and comparing the women in the intervention clinics for whom the clinical care path was actually used to all other women (both those who were at an intervention clinic but did not receive the clinical care path and those in the control group); 2) comparing results in women with and without complete data.

Investigators will perform subgroup analysis to examine the outcomes at obstetrician clinics separately from those at midwifery clinics. Potential covariates which may not be evenly distributed between the intervention and control groups will be controlled for (e.g. age, socioeconomic status, etc). Since observations within each participating clinic will be assumed more likely to be similar than observations between clinics, a logistic model using a conditional (for paired data) generalized estimating equation (GEE) method will be performed to account for this clustering effect within clinics, incorporating both within-clinic and between-clinic variations. An intracluster correlation coefficient (ICC) and variance inflation factor (VIF) will also be calculated to assess the impact of the clustering effect.

Results will be considered statistically significant at two-sided alpha=0.05 . A modified Bonferroni correction will be used given the multiple secondary outcomes. Analyses will be performed using SAS-PC statistical software (version 9.2; SAS institute Inc, Cary, NC).

TEAM:

Principal Investigator: Sarah McDonald, MD, MSc (Clinical Epidemiology), is an obstetrician and Associate Professor, McMaster University and Tier II Canada Research Chair in Maternal and Child Obesity Prevention and Intervention. Maternal weight and weight gain are the focus of her research program. She will oversee all aspects of this study.

Co-Investigators:

Lucy Giglia, MD, MSc (Epidemiology), a pediatrician, Associate Clinical Professor, McMaster University and a former Health Canada epidemiologist, is the Research Lead for the Division of General Pediatrics at McMaster Children's Hospital.

Lehana Thabane, PhD, a statistician/RCT expert, is the Associate Chair of the Department of Clinical Epidemiology and Biostatistics and the Director of the Biostatistics Unit at the Centre for Evaluation Medicine, McMaster University and is experienced in the design, management and analysis of both RCTs and pilot RCTs.

Collaborator:

Cindy Maxwell, MD, was the co-author on the national guideline on the care of obese pregnant women, and the head of an obesity clinic for pregnant women at Mount Sinai Hospital in Toronto.

Clinicians whose clinics would be potential recruitment sites have been and will continue to be involved in all phases of the study and development of the care pathway.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for clinics:

  1. location in southwestern Ontario (for proximity to the research team),
  2. availability of a clinician willing to serve as the local site lead, and
  3. lack of any type of existing clinical care pathway for obese pregnant women
* Inclusion criteria for participants:

  1. women with a pre-pregnancy (or in the event of inability to recall, then first measured) BMI >30 kg/m2
  2. with viable singleton pregnancies up to 20 weeks + 6 days gestational age upon first visit to randomized clinic

Exclusion Criteria:

* Women with:

  1. a miscarriage or termination of pregnancy after enrollment,
  2. twins or higher order multiples or
  3. a fetus with a known lethal anomaly.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2015-10; Primary Completion 2017-04-30 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility (Rates) | 10 months
  1. the feasibility of the intervention (defined as >80%: A. compliance with each step in care path and B. clinicians recommend it.)
  2. the feasibility of a cluster RCT (defined as >80%: A. randomization (of approached clinics), B. uptake (of eligible women), C. completeness of follow-up.

SECONDARY OUTCOMES:
Process outcome - Rates of offer | 10 months
  1. T1: rates of offer of testing for pre-existing diabetes with 75g OGTT or 50g GCT, nuchal translucency u/s, calculation of body mass index, BMI, counselling about weight gain, advising about medical complications, screening for obstructive sleep apnea, referral to maternal-fetal medicine if history of bariatric surgery,
  2. T2: offer of maternal-serum alpha fetal protein testing for spina bifida, anatomy ultrasound, and 50g GCT and 75g OGTT,
  3. T3: offer of consultation with anaesthesiology, ultrasound for growth & wellbeing, counselling for risk of operative vaginal delivery, shoulder dystocia, caesarean section, and discussion of breastfeeding.
  Prior to data collection, due to feasibility issues, we focused Carepath use to the antenatal period.
Exploratory clinical outcomes - Rates of detection | 10 months
  Fetal abnormalities:
  1. cardiac,
  2. neural tube or
  3. other defects.
  Maternal outcomes:
  1. type 2 diabetes,
  2. gestational diabetes,
  3. sleep apnea.
Provider outcomes - Questionnaire --Rates of | 10 months
  1. acceptability (defined as >80% would recommend it to a colleague)
  2. feasibility (defined as >80% found it easily accomplished during routine care)
  3. usefulness (defined as >80% thought women more likely to receive appropriate care with it)
  4. barriers and facilitators to the intervention; mechanisms or factors that impact its ease of use and effectiveness and for its improvement (through structured interviews, the questions for which have been drafted)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah D McDonald, MD, MSc, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada